CLINICAL TRIAL: NCT04502238
Title: Dehydration and Population Health
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Wayne State University (Other)
Collaborators: University of Chicago (Other)
Responsible Party: Principal Investigator, Tamara Hew-Butler DPM, PhD, FACSM, Associate Professor, Exercise and Sport Science, Wayne State University
Other Study IDs: 1908002467
Record Dates: First submitted 2020-07-28; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Dehydration (Physiology)
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fluid restriction — Study participants will refrain from drinking fluids overnight to facilitate 1-2% fluid loss from baseline

SUMMARY:
The primary aim of this study is to assess cardiovascular changes (blood pressure, heart rate, electrocardiogram/ECG) in response to mild fluid-restriction dehydration and subsequent rehydration in healthy young and old people. Secondary aims are to assess changes in body composition, mood, and hunger in response to mild dehydration and rehydration.

DETAILED DESCRIPTION:
PARTICIPANTS: Forty healthy (no regular prescription medication use) male and females, between the ages of 18-70 years, will be recruited for this randomized-control cross-over study. Ideally, the investigators hope to recruit twenty "younger" (18-50) and twenty "older" (50-70) participants for this pilot study.

All participants will be required to participate in two separate trials (a control and dehydration-rehydration trial, in randomized order), separated by at least a week. All menstruating females will be tested during the follicular phase of their menstrual cycle (i.e. within the first 14 days after the onset of the menstrual period). All participants will present to the lab in the evening for pre-testing and then in the morning for mid-testing/post-testing. With both pre-testing and mid-testing/post-testing each taking ~90 minutes each, plus 12-hours of fluid deprivation or regular food/fluid intake overnight, the total time participating in collective study activities would be approximately 30-hours (~15 hours per trial).

PROCEDURES: For each of the two study trials, participants will come to the lab in the evening for pre-testing and then the following morning for mid-testing/post-testing (one trial). Hydration status will be assessed using blood (venipuncture), urine (spot sample), body weight, and thirst rating (100mm visual analogue scale). Cardiovascular variables will be assessed via heart rate, ECG, and blood pressure. Body composition will be measured using a dual energy x-ray absorptiometry (DXA) scan. Mood will be assessed using the Profile of Mood States (POMS) questionnaire.

Once the participants present to the lab, pre-test blood, urine, body weight and composition, mood and thirst/sodium/hunger ratings will be obtained. Then, to enhance sweat water losses, each participant will be asked to walk on a motorized treadmill at a self-selected speed for 60-minutes.

During the Dehydration-Rehydration trial, participants will be asked to refrain from ingesting any fluid (fluid restriction) for at least 12-hours overnight (i.e. from leaving the lab that evening until coming into the lab the next morning) to facilitate dehydration. After mid-testing, the participants will be allowed free access to water for a 60-minute rehydration period to quench their thirst ("ad libitum" drinking). At the end of this 60-minute rehydration period, post-test measures will be repeated. During the control trial, the participants can eat and drink as they please during the 12-hour overnight period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (no regular prescription medication usage)
* Able to walk continuously on treadmill for 60 minutes

Exclusion Criteria:

* Confirmed or suspected pregnancy
* Chronic medical condition
* Regular prescription medication use
* Inability to walk continuously walk on a treadmill for 60 minutes

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy (i.e. does not take any regular prescription medications) adults between the ages of 18-70 years, who can walk comfortably on a treadmill for 1-hour (to enhance fluid loss before the rehydration period).
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-11-06 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular changes | change from baseline to dehydration (+13 hours) and then rehydration (+15 hours)
  Changes in QRS waveforms will be assessed using electrocardiograms (ECG) before and after dehydration (fluid restriction)

SECONDARY OUTCOMES:
Changes in perception of thirst and hunger | change from baseline to dehydration (+13 hours) and then rehydration (+15 hours)
  Thirst and hunger will be assessed on a VAS (visual analogue scale) before and after dehydration (fluid restriction)
Changes in body composition | change from baseline to dehydration (+13 hours) and then rehydration (+15 hours)
  Body composition (bone, lean, and fat mass) will be assessed using dual energy x-ray absorptiometry (DXA) scans before and after dehydration (fluid restriction)
Changes in mood | change from baseline to dehydration (+13 hours) and then rehydration (+15 hours)
  Mood will be assessed using the POMS (profile of mood states) survey before and after dehydration (fluid restriction)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara D Hew(-Butler), PhD, Principal Investigator — Wayne State University
Locations (1):
- #055 Education Building, Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
All data shared, especially with regards to our University of Chicago collaborators, will be de-identified. Participants will be assigned an unidentified subject number once consent form is signed, and all data collected and imported into a spreadsheet will be de-identified. The "master list" which contains the link between each participant's name and the assigned subject number will be placed in a locked cabinet in Dr Hew-Butler's office, separate from the actual data and signed informed Consent forms. All participant information will remain strictly confidential and will not be identified in any subsequent publications or presentation of the results.